CLINICAL TRIAL: NCT04615156
Title: Evaluation of 18F-2-fluoro-2-deoxy-D-glucose Produced by a New Manufacturer, for Safety, Through the Identification of Adverse Events, and Efficacy, Through the Evaluation of Its Ability, When Utilized in Performance of a Positron Emission Tomography Computed Tomography Scan, to Correctly Distinguish Benign From Malignant Solitary Pulmonary Nodules.
Brief Title: 18F-2-fluoro-2-deoxy-D-glucose in Positron Emission Tomography Computed Tomography
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eastern Health, Canada (Other)
Responsible Party: Principal Investigator, Dr. Jeffery Flemming, Clinical Chief, Nuclear and Molecular Medicine, Eastern Health, Eastern Health, Canada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 231364; 231364 (Other: Protocol number assigned by Health Canada)
Record Dates: First submitted 2020-10-28; First posted 2020-11-04 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Solitary Pulmonary Nodule; Oncology; 18F-2-fluoro-2-deoxy-D-glucose; Adverse Event
Keywords: 18F-2-fluoro-2-deoxy-D-glucose; Adverse Event; Solitary Pulmonary Nodule; Oncology
MeSH Terms: conditions — Solitary Pulmonary Nodule; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation for adverse events from 18F-2-fluoro-2-deoxy-D-glucose produced by a new manufacturer (Experimental)
  Interventions: Drug: 18F-2-fluoro-2-deoxy-D-glucose

INTERVENTIONS:
Drug: 18F-2-fluoro-2-deoxy-D-glucose — Administration of 18F-2-fluoro-2-deoxy-D-glucose for the purposes of diagnosis.

SUMMARY:
The study objectives are as follows:

* To determine the safety of trial 18F-2-fluoro-2-deoxy-D-glucose, produced by a new manufacturer, by surveillance for adverse events in patients having Positron Emission Tomography Computed Tomography scans in a comprehensive program for indications including, but not limited to, oncology, neurology, cardiac and infectious/inflammatory processes.
* To determine the efficacy of 18F-2-fluoro-2-deoxy-D-glucose Positron Emission Tomography in differentiating benign from malignant solitary pulmonary nodules and calculate sensitivity, specificity, and accuracy using pathologic confirmation as the gold standard when available, or greater than 6 month follow up stability on Computed Tomography scan when not.

The purpose of performing this clinical trial is to provide local access of 18F-2-fluoro-2-deoxy-D-glucose to the patients of Newfoundland and Labrador. This product has been offered to patients over the last three years by transporting from facilities outside of the province. There have been significant delays in access and in fact, times where 18F-2-fluoro-2-deoxy-D-glucose has not been available through this process. This has caused delays and limitations of treatments for patients who rely on Positron Emission Tomography Computed Tomography scans for diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Known or suspected disease for which 18F-2-fluoro-2-deoxy-D-glucose Positron Emission Tomography Computed Tomography is appropriate for the investigation of. This includes, but is not limited to: Known or suspected cancer, neurological disorders (dementia or epilepsy), cardiac conditions (inflammation or myocardial viability), known or suspected presence of infection/inflammation process

Patients must satisfy all the following:

* Able to provide written informed consent, or consent obtained from appropriate guardian
* Able to tolerate the physical and logistic requirements of completing a Positron Emission Tomography Computed Tomography scan

Exclusion Criteria:

* Pregnant women: if there is any possibility of pregnancy, a blood Beta Human Chorionic Gonadotropin level will be obtained as per Eastern Health policy.
* Patients unwilling or unable to stop breast feeding for 12 hours
* Patients who are too medically unstable to tolerate the uptake period or lie flat for the duration of the scan
* Patients who exceed the safe weight limit of the Positron Emission Tomography Computed Tomography scanner bed (500 lbs.) or who cannot fit through the bore (70 cm diameter)
* Patients unwilling to proceed with scan (I.e. claustrophobia) prior to injection
* If patients inability to follow staff direction causes a safety hazard prior to injection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2020-11-01 (Estimated); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Measuring the safety of 18F-2-fluoro-2-deoxy-D-glucose produced by a new manufacturer by evaluating for any adverse events that occur during their Positron Emission Tomography Computed Tomography scan appointment. | For the length of time required to perform informed consent, the scan, and follow-up interview for adverse events, approximately 4 hours
  Evaluation for any adverse events after administration of 18F-2-fluoro-2-deoxy-D-glucose produced by Eastern Health in the Nuclear and Molecular Medicine Department who is a new manufacturer

SECONDARY OUTCOMES:
Evaluation of the sensitivity, specificity and accuracy of 18F-2-fluoro-2-deoxy-D-glucose in the assessment of solitary pulmonary nodules compared to anatomic pathology, or more than 6 month follow-up stability when not available. | Variable, from the time of the scan to appropriate follow-up (either biopsy or follow-up imaging that occurs more than 6 months after the Positron Emission Tomography Computed Tomography study)
  Assess the sensitivity, specificity and accuracy of 18F-2-fluoro-2-deoxy-D-glucose Positron Emission Tomography Computed Tomography in differentiating benign from malignant solitary pulmonary nodules. This is being done with a view towards eventually applying for an Abbreviated New Drug Submission.

IPD SHARING:
Plan to Share IPD: No